CLINICAL TRIAL: NCT07008456
Title: A Phase II Study to Investigate the Efficacy and Safety of Two Different Doses of Twice Daily Distal Jejunal-release Dextrose Beads Formulations (APHD 012 and APHD 002) Combined With a Gel Composition, Compared With Two Different Doses of the Placebo Beads Formulations (APHP 012 and APHP 002) Combined With a Gel Composition in Obese Subjects With Weight Related Comorbidities
Brief Title: A Study to Investigate the Efficacy and Safety of Two Different Doses of Twice Daily Distal Jejunal-release Dextrose Beads Formulations Combined With a Gel Composition Compared to Placebos in Obese Subjects With Weight Related Comorbidities
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aphaia Pharma US LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AP2501
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Obese With Comorbidities; Obese Patients (BMI ≥ 30 kg/m²)
Keywords: obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- APHD-012 (Active Comparator): 12 g dextrose beads
  Interventions: Drug: APHD-012
- APHD-002 (Active Comparator): 2 g dextrose beads
  Interventions: Drug: APHD-002
- APHP-012 (Placebo Comparator): 12 g placebo beads
  Interventions: Drug: APHP-012
- APHP-002 (Placebo Comparator): 2 g placebo beads
  Interventions: Drug: APHP-002

INTERVENTIONS:
Drug: APHD-012 — 12 g dextrose beads
  Arms: APHD-012
Drug: APHD-002 — 2 g dextrose beads
  Arms: APHD-002
Drug: APHP-012 — 12 g placebo beads
  Arms: APHP-012
Drug: APHP-002 — 2 g placebo beads
  Arms: APHP-002

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled, phase IIa study is to demonstrate superiority on body weight reduction of two different doses of twice daily distal jejunal-release dextrose beads formulations (APHD 012 and APHD 002) combined with a gel composition, compared with two different doses of the placebo beads formulations (APHP 012 and APHD 002) combined with a gel composition in obese subjects with weight related comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between an age of 18 (or the legal age of consent in the jurisdiction where the study is conducted) and 75 at the time of signing Informed Consent Form (ICF).

  2. Body Mass Index (BMI) of
  1. ≥30 kg/m2
  2. ≥27 kg/m2 and <30 kg/m2 with at least 1 of the following weight-related comorbidities

     * hypertension: on blood-pressure (BP)-lowering medication or having systolic BP (SBP) ≥140 mmHg or diastolic BP (DBP) ≥90 mmHg at Screening
     * dyslipidaemia: on lipid-lowering medication or having low-density lipoprotein (LDL) ≥160 mg/dL (4.1 mmol/L) or triglycerides ≥150 mg/dL (1.7 mmol/L), or high-density lipoprotein (HDL) <40 mg/dL (1.0 mmol/L) for men or HDL <50 mg/dL (1.3 mmol/L) for women at Screening
     * cardiovascular disease (for example, ischemic cardiovascular disease, New York Heart Association [NYHA] Functional Classification Class I-II heart failure.)
     * obstructive sleep apnoea (only in participants >30 years of age) 3. Stable body weight for the 3 months prior to randomization (<5% body weight gain and/or loss) 4. History of at least one self-reported unsuccessful dietary effort to lose body weight 5. Fully vaccinated against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) during Coronavirus Disease 2019 (COVID-19) pandemic. Full Vaccination means having received all recommended doses of a COVID-19 vaccine listed by either of World Health Organization (WHO)-Emergency Use Listing (WHO-EUL), Food and Drug Administration (FDA) or European Medicines Agency (EMA) or a mix and match series composed of any heterologous combination of WHO-EUL/FDA/EMA-approved or authorized COVID-19 vaccines. Alternatively, a proven recovery from a COVID-19 infection in combination with at least one vaccination with a WHO, FDA, EMA listed vaccine qualifies as a full vaccination. The vaccination program must have been completed at least two weeks prior ICF signed. For the avoidance of doubt, the vaccination scheme received shall be in compliance with the current rules defined by the relevant health authorities in the US or Europe.

       6. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol

     Exclusion Criteria:
* 1. Prior or planned surgical treatment for obesity (excluding liposuction or abdominoplasty, if performed >1 year prior to screening) 2. Obesity induced by other endocrinologic disorders (for example, Cushing's syndrome) or diagnosed monogenetic or syndromic forms of obesity (for example, Melanocortin 4 Receptor deficiency or Prader-Willi Syndrome) 3. Plan to have endoscopic and/or device-based therapy for obesity or have had device removal within the last 12 months prior to screening including but not limited to

  * mucosal ablation
  * gastric artery embolization
  * intragastric balloon
  * duodenal-jejunal endoluminal liner. 4. Renal impairment measured as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 during screening.

    5. Any of the following: myocardial infarction, stroke, hospitalization for unstable angina or transient ischaemic attack within the past 60 days prior to screening 6. Subject presently classified as being in New York Heart Association (NYHA) Class III and IV 7. Elevated resting pulse rate (>100 bpm) at Screening and Visit 1 8. Electrocardiogram (ECG) considered clinic ally significant by the Investigator at Screening 9. Known clinically significant gastric emptying abnormalities (for example, severe gastroparesis or gastric outlet obstruction), past gastric bypass (bariatric) surgery or restrictive bariatric surgery (for example, Lap-Band®), or chronic intake of drugs directly affecting gastrointestinal (GI) motility 10. History or presence of acute or chronic pancreatitis. 11. History or presence of acute or chronic diverticulitis or diverticulosis. 12. History or presence of a clinically significant active autoimmune abnormality (for example, lupus or rheumatoid arthritis) 13. History or presence of clinically significant gallbladder disease 14. Signs and symptoms of any other liver disease other than non-alcoholic fatty liver disease, or any of the following as determined during screening
  * Alanine aminotransferase (ALT) level >3.0X Upper limit of normal (ULN) for the reference range
  * Alkaline phosphatase (ALP) level >1.5X ULN for the reference range, or
  * Total Bilirubin >1.5X ULN for the reference range (except for cases of known Gilbert's Syndrome) 15. Evidence of hypothyroidism or hyperthyroidism based on clinical evaluation and/or an abnormal thyroid-stimulating hormone that, in the opinion of the Investigator, would pose a risk to patient safety. Subjects on a stable dose of thyroid replacement therapy for at least the prior 3 months before Visit 1 who are clinically euthyroid and who are anticipated to remain on this dose throughout the trial period may be eligible if they meet the other criteria 16. Known self or family history (first-degree relative) of multiple endocrine neoplasia type 2A or type 2B, thyroid C-cell hyperplasia, or medullary thyroid carcinoma 17. Eating habits consisting of eating relevant amounts of food throughout the night (after 10 p.m.; except if working on night shifts) 18. History or presence of bulimia or anorexia nervosa 19. History or presence of significant active or unstable Major Depressive Disorder (MDD) or other severe psychiatric disorder (for example, schizophrenia, bipolar disorder, or other serious mood or anxiety disorder) within the last 2 years.

    20. Lifetime history of suicide attempt 21. History of malignant neoplasms within the past 5 years prior to screening. Basal and squamous cell skin cancer and any carcinoma in-situ are allowed 22. Evidence of human immunodeficiency virus (HIV) and/or positive HIV antibodies historically or at Screening 23. Evidence of hepatitis B and/or positive hepatitis B surface antigen. 24. Hepatitis C as defined by presence of positive hepatitis C antibodies. 25. Unstable treatment with glucose-lowering agent(s) within 90 days before Visit 1 26. Treatment with incretin mono- or dual receptor agonists (e.g., Glucagon-like peptide 1 (GLP-1) or GLP-1/ Glucose-dependent insulinotropic polypeptide (GIP)) within 180 days prior to screening and planned during the present study 27. Use of non-herbal Chinese medicine or other non-herbal local medicine with unknown/unspecified content within 90 days before screening 28. Surgery scheduled for the duration of the trial, except for minor surgical procedures, in the opinion of the investigator 29. Known or suspected abuse of alcohol or recreational drugs 30. Illicit drug abuse (marihuana, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines) 31. Known or suspected hypersensitivity to trial product(s) or related products 32. Participation in another clinical trial within 90 days before screening 33. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method 34. Any disorder, unwillingness or inability, not covered by any of the other exclusion criteria, which in the investigator's opinion, might jeopardize the subject's safety or compliance with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Body weight | 24 weeks
  Mean percent change in body weight from Baseline at Week 24

SECONDARY OUTCOMES:
Blood Pressure | 24 weeks
  Change in blood pressure (systolic and diastolic blood pressure) from Baseline at Week 24
Lipoproteins lipids | 24 weeks
  Change in lipoprotein lipids (Low-density lipoprotein cholesterol (LDL-C) and High-density lipoprotein cholesterol (HDL-C) from Baseline at Week 24
Fasting Glucose | 24 weeks
  Change in fasting glucose from Baseline at Week 24
HbA1c | 24 weeks
  Change in HbA1c (in subjects with Type 2 Diabetes Mellitus) at Week 24

CONTACTS AND LOCATIONS:
Locations (6):
- Georgia (6):
  - LTD "Israeli-Georgian Medical Research Clinic Healthycore", Tbilisi, K'alak'i T'bilisi
  - LTD "New Hospitals", Tbilisi, K'alak'i T'bilisi
  - LTD "Acad. G. Chapidze Emergency Cardiology Center", Tbilisi, K'alak'i T'bilisi
  - LTD "Diacor", Tbilisi, K'alak'i T'bilisi
  - NNLE "Jo Ann University Hospital", Tbilisi, K'alak'i T'bilisi
  - LTD The First Medical Center, Tbilisi, K'alak'i T'bilisi

IPD SHARING:
Plan to Share IPD: Undecided